CLINICAL TRIAL: NCT07144371
Title: Effects of Virtual Reality-based Cognitive and Technical Drills on Scanning and Passing Performance in Youth Football Players: a Randomized Controlled Study
Brief Title: VR-Based Cognitive & Technical Training in Youth Football: A Randomized Trial
Acronym: VR-SCANPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Sağlık ve Teknoloji Üniversitesi (Other)
Responsible Party: Principal Investigator, Sena Çınarlı, Ass Prof, Kocaeli Sağlık ve Teknoloji Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ES-VR-01
Record Dates: First submitted 2025-08-17; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2023-02

CONDITIONS: Virtual Reality; Football; Training Study; Cognitive Performance
Keywords: cognitive training; scanning behavior; passing performance; perceptual skills
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This study used a parallel-group, randomized controlled design. Twenty-two youth football players (U16-U17) were randomly allocated to either a Virtual Reality (VR) training group or a Control group (n = 11 per group). The intervention lasted 7 weeks, with three VR training sessions per week in addition to regular football practice. The Control group continued regular football training only. Outcomes included scanning frequency and passing performance assessed during structured small-sided games.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Training Group (Experimental): Participants in this arm completed a 7-week virtual reality training program in addition to their regular football practice. The VR training was performed three times per week using the SensiballVR™ system, which integrates immersive cognitive drills (multi-object tracking, peripheral vision, scanning tasks) with football-specific technical passing scenarios under time pressure.
  Interventions: Other: Virtual Reality Training Group
- Control Group (Active Comparator): Participants in this arm continued their regular football training sessions over the 7-week period. They did not receive any additional VR-based training. This group served as the control condition for comparison with the experimental VR group.
  Interventions: Other: Standard Football Training

INTERVENTIONS:
Other: Virtual Reality Training Group — Participants continued their routine football training program with no additional VR-based training. This group served as the active comparator to evaluate the relative effects of VR training on scanning frequency and passing performance.
  Other Names: Control Group
  Arms: Virtual Reality Training Group
Other: Standard Football Training — Participants continued their routine football training program with no additional VR-based training. This group served as the active comparator to evaluate the relative effects of VR training on scanning frequency and passing performance.
  Arms: Control Group

SUMMARY:
In recent years, virtual reality (VR) has emerged as a promising tool to bridge this gap. By providing immersive, interactive, and customizable environments, VR-based interventions offer a safe and controlled platform for simulating complex game scenarios (7). From a neurophysiological perspective, VR training can stimulate the activation of key brain regions involved in perception, attention, and decision-making (8). Recent research examined the relationship between perceptual-cognitive performance in a dynamic 360° environment and soccer-specific performance in youth players (9). Their findings indicated a significant positive correlation between performance in a 360° multiple object tracking task and both passing accuracy and defensive effectiveness in small-sided games.

The repeated exposure to dynamic, visually rich stimuli enhances selective attention, working memory, and anticipatory skills, which are all critical for effective environmental scanning (10,11). Furthermore, the real-time feedback and motor engagement involved in VR-based drills promote sensorimotor integration, strengthening the neural pathways that support technical execution, such as passing accuracy and timing (12). These findings suggest that VR is not merely a visual aid but a cognitive training modality capable of eliciting measurable changes in sport-specific decision-making and technical performance (13).

However, current literature is still limited in terms of randomized controlled trials investigating the combined effects of VR on scanning and passing performance in football players. Therefore, this study aimed to evaluate the effects of a VR-based training program that integrates cognitive and technical drills on scanning behavior and passing performance in youth footballers. It was hypothesized that VR-based training intervention would demonstrate significantly greater improvements in scanning frequency and passing accuracy compared to those in the control group receiving only traditional training.

DETAILED DESCRIPTION:
The present parallel-group randomized controlled trial was designed to investigate the effects of a 7-week VR-based training program on scanning behavior and passing performance in youth football players. A total of 22 male athletes from U16-U17 categories were recruited from a regional football academy. Inclusion criteria required participants to be injury-free in the last 12 months, possess normal or corrected-to-normal vision, and have no prior exposure to VR training. Players with neurological or vestibular disorders, or recent orthopedic surgery, were excluded. Participants and their legal guardians provided informed consent prior to participation.

Participants were randomly assigned (1:1) to either the VR training group (n = 11) or a control group (n = 11). Randomization was stratified by age and playing position to ensure group equivalence. The control group continued their regular football training program, while the VR group participated in an additional VR training intervention delivered via the SensiballVR™ platform three times per week for seven weeks (21 sessions in total). Each VR session targeted two core domains: (1) scanning frequency through tasks requiring frequent and purposeful exploration of the virtual pitch, and (2) technical passing performance through drills simulating teammate and opponent interactions under time pressure. The VR system incorporated HTC Vive Pro Eye headsets and patented haptic footwear technology, providing tactile feedback and precise motion tracking to ensure ecological validity. Training intensity was progressively increased across three phases, from basic visual exploration to advanced dual-task drills with complex passing demands.

Outcome measures included (a) scanning frequency classified as before ball reception, during control, and off-the-ball actions, and (b) passing performance categorized by execution type (one-touch, control-pass, multi-touch), outcome (successful or unsuccessful), and style (short, penetrative, long). All data were collected during structured small-sided games (5v5+1 and 7v7+7 joker formats) and analyzed via synchronized aerial and ground-level video recordings. Notational analysis was conducted by two independent analysts with excellent inter-rater reliability (ICC > 0.90).

Statistical analyses were performed using non-parametric tests due to violations of normality in several variables. Within-group changes were assessed using the Wilcoxon signed-rank test, while between-group comparisons of delta scores (post-pre) were evaluated using the Mann-Whitney U test. Effect sizes (r) were calculated and interpreted using conventional thresholds. Percentage changes in mean values were also reported to illustrate practical relevance.

ELIGIBILITY:
Inclusion Criteria:

* Male youth football players (U16-U17 age categories)
* Injury-free in the past 12 months
* Normal or corrected-to-normal vision
* No prior exposure to virtual reality-based training

Exclusion Criteria:

* Presence of neurological disorders
* Presence of vestibular disorders
* History of recent orthopedic surgery

Ages: 16 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Scanning Frequency in Small-Sided Games | Baseline (pre-intervention) and after 7 weeks of training
  Scanning behavior will be assessed during structured small-sided games and categorized into three domains: (1) before ball reception, (2) during ball control, and (3) off-the-ball. Each scanning action will be coded from synchronized video recordings by trained analysts using standardized operational definitions. Outcomes will be expressed as the number of scanning actions per game and analyzed for changes from baseline to post-intervention.

SECONDARY OUTCOMES:
One-Touch Short-Successful Passes | Baseline and after 7 weeks of training
  Number of short passes executed successfully with one touch during small-sided games. Passes will be coded from synchronized video analysis using predefined operational criteria.
Control-Pass Short-Successful Passes | Baseline and after 7 weeks of training
  Number of short passes executed successfully following initial ball control (≥2 touches not allowed). Actions will be coded via video analysis by two trained observers.
Penetrative-Successful Passes | Baseline and after 7 weeks of training
  Number of successful deep passes that eliminate at least two opponents before reaching a teammate. Includes one-touch and control-pass executions.
Long-Successful Passes | Baseline and after 7 weeks of training
  Number of successful aerial (long) passes delivered to a teammate. Includes one-touch and control-pass executions.
Passing Efficiency | Baseline and after 7 weeks of training
  Ratio of successful passes to total passes executed during small-sided games. All pass types (one-touch, control, multi-touch) will be included.

CONTACTS AND LOCATIONS:
Locations (1):
- Eskişehir Technical University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have not yet determined whether individual participant data (IPD) will be shared.

REFERENCES:
- [Background] Lachowicz M, Zurek A, Jamro D, Serweta-Pawlik A, Zurek G. Changes in concentration performance and alternating attention after short-term virtual reality training in E-athletes: a pilot study. Sci Rep. 2024 Apr 17;14(1):8904. doi: 10.1038/s41598-024-59539-w. PMID 38632364
- [Derived] Erisik K, Cerrah AO, Cinarli FS. Effects of virtual reality-based cognitive and technical drills on scanning and passing performance in youth football players: a randomized controlled study. BMC Sports Sci Med Rehabil. 2025 Dec 24;17(1):371. doi: 10.1186/s13102-025-01425-7. PMID 41444702